CLINICAL TRIAL: NCT03576339
Title: Influence of Electrical Stimulation on Palatal Wound Healing. Randomized Clinical Trial
Brief Title: Influence of Electrical Stimulation on Palatal Wound Healing.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Assistant professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UEPJMF9
Record Dates: First submitted 2018-06-05; First posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Palatal Wound
Keywords: Wound Healing; Electrical Stimulation; Palatal
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Group - Free Gingival Graft + Sham Electric Stimulation (Sham Comparator): With the aim to ridge preservation after condemned tooth extraction, the socket will be sealed with a free gingival graft removed from the palate. The tooth will be extracted through the use of appropriate instruments in order to obtain a minimally traumatic exodontia. After the exodontia, curettage and irrigation of the dental socket will be performed. The free gingival graft will be removed from the donor palatal area with a circular incision of 9 mm and 2 mm thickness. After free gingival graft removal from palate, it will be adjusted to the entrance of the socket and sutured. Patient randomized to the SHAW Group will receive the simulation of the electrical stimulation process, thus non current will be applied.
  Interventions: Procedure: Free Gingival Graft; Device: SHAM Electric stimulation
- Test Group - Free Gingival Graft + Electric Stimulation (Experimental): With the aim to ridge preservation after condemned tooth extraction, the socket will be sealed with a free gingival graft removed from the palate. The tooth will be extracted through the use of appropriate instruments in order to obtain a minimally traumatic exodontia. After the exodontia, curettage and irrigation of the dental socket will be performed. The free gingival graft will be removed from the donor palatal area with a circular incision of 9 mm and 2 mm thickness. After free gingival graft removal from palate, it will be adjusted to the entrance of the socket and sutured. Conductive electrodes for electrical current application will be applied to the palatal donor area on each side of the wound at a distance of 3 mm from the wound edge. An alternating current of 100 microamperes (μA) at 9 kilohertz (kHz), will be distributed in order to traverse the operated area. A single application of electrical stimulation will be given for 120 seconds, five consecutive days.
  Interventions: Procedure: Free Gingival Graft; Device: Electric Stimulation

INTERVENTIONS:
Procedure: Free Gingival Graft — Free gingival graft removal from palate for socket preservation
  Other Names: Socket preservation
Device: SHAM Electric stimulation — Simulation of electric stimulation protocol for 120 seconds once a day in five consecutive days. In Sham stimulation non current will be applied.
  Arms: Sham Group - Free Gingival Graft + Sham Electric Stimulation
Device: Electric Stimulation — Local Electric Stimulation for 120 seconds once a day in five consecutive days.
  Other Names: Local Electric Stimulation
  Arms: Test Group - Free Gingival Graft + Electric Stimulation

SUMMARY:
The aim of this present study is to evaluate the clinical and patients-centered parameters of electric stimulation on wound healing process of the donor palatal area after free gingival graft (FGG) removal.

DETAILED DESCRIPTION:
This is a randomized, parallel, double-blind clinical trial. The population that will be evaluated in this is study will be select at Science and Technology Institute - ICT-Sao Jose dos Campos, College of Dentistry.

Patients will be assigned to one of the treatments groups:

* Sham Group - Free Gingival Graft (n = 22): Atraumatic extraction surgery and free gingival graft for sealing the entrance of the alveolus associated with SHAM electrical stimulation simulation.
* Test Group - Free Gingival Graft + Electric stimulus (n = 22): Atraumatic extraction surgery with placement of a free gingival graft to seal the entrance of the alveolus associated with electrical stimulation in the open wound on the palate.

All surgeries will be performed by the same expert periodontist (MMVM). A blade 15c (Swann-Morton® - Sheffield, England) mounted on No. 3 scalpel handle will make an intrasulcular incision around the tooth indicated for exodontia. Then, the tooth will be extracted through the use of appropriate instruments in order to obtain a minimally traumatic exodontia. With the aim to ridge preservation after tooth extraction the socket will be sealed with a free gingival graft removed from the palate. For the free gingival graft removal, a circular template of 9 millimeters in diameter will be used. This mold has the objective of standardizing the palatal graft removal ensuring the wounds will have always the same size. After the circular incision, the graft will be removed with a thickness of 2 millimeters. After free gingival graft removal from palate, it will be adjusted to the entrance of the socket and sutured with Vicryl® 5.0 reabsorbable (Ethicon Johnsons do Brasil, São José dos Campos - SP).

For electrical stimulation, a unit consisting of a signal generator (Keysight Technologies., Inc., Santa Rosa-CA, USA), a power supply (Keysight Technologies., Inc., Santa Rosa-CA, USA) and circuit board will be used. Conductive electrodes for electrical current application will be applied to the palatal donor area on each side of the wound at a distance of 3 mm from the wound edge. An alternating current of 100 microamperes (μA) at 9 kilohertz (kHz), will be distributed in order to traverse the operated area. A single application of electrical stimulation will be given for 120 seconds, five consecutive days. The electric current will have its visualization optimized through an oscilloscope. Patients randomized to the Control Group (SHAM) will receive the simulation of the electrical stimulation (ES) process.

The evaluated clinical parameters will be: wound remaining area (WRA), scar and tissue colorimetry (TC), tissue thickness (TT) and epithelization (E). Moreover, patient-centered also will be evaluated as: number of pills (NP), tissue edema (TE), postoperative discomfort (D) and Oral Health Impact Profile (OHIP).

All data will be expressed as mean ± standard deviation (SD), and normality will be tested using the Shapiro-Wilk test. Values for remaining wound area, scar and tissue colorimetry, tissue thickness, and epithelization will be examined by repeated measures ANOVA to assess differences within and between groups, followed by a Tukey test for multiple comparisons when the value of p Shapiro-Wilk ≥ 0.05. Those with Shapiro-Wilk p values <0.05 will be analyzed using the Friedman test (for intragroup comparisons) and Mann-Whitney tests (for intergroup comparisons). Values referring to patient-centered parameters such as postoperative discomfort, the number of analgesics taken, tissue edema and oral health impact profile measurements will be analyzed using the T-Test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 18 years of age, systemically healthy, with good oral hygiene, assessed by plaque index and gingival index of less than 25% (O'Leary et al., 1972);
* Patients with no morphological or pathological changes in the donor palatine region;
* Patients who present indication of exodontia and with ridge preservation indication for future implantation of implants;
* The tooth included in the study, as well as the adjacent teeth do not present a loss of periodontal insertion;
* Patients who agreed to and signed the formal consent to participate in the study after receiving an explanation of risks and benefits from an individual who was not a member of the present study (Resolution no. 118 - May, 2012, and Ethics and Code of Professional Conduct in Dentistry - 118/12).

Exclusion Criteria:

* Patients with systemic problems (cardiovascular, blood dyscrasias, immunodeficiency, and diabetes, among others) that will contraindicate the surgical procedure;
* Patients taking medications known to interfere with the wound healing process or that contraindicate the surgical procedure;
* Smokers patients;
* Pregnant or lactating patients;
* Patients who had had periodontal surgery on the study area;
* Patients who present opportunistic oral lesions, mainly colonized the palate region;
* Patient using a pacemaker.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Remaining wound area | 7 days
  The defect area will be measured after 7 post-operative days. For this, standardized photography will be taken ( in terms of brightness, distance and angle). A scale will be used as a reference to measure the area. These photographs will be exported to image software (Image J-NIH, Bethesda, USA) and the wound area will be measured in square millimeters (mm2) (Dias et al. 2015).

SECONDARY OUTCOMES:
Scar and tissue colorimetry | 30 days
  Will be analyzed presence or absence of scar in the operated area after 30 days post-operative. Moreover, Tissue color similarity between the region adjacent to the operated area and the post-operative image were analyzed through photographs. The photographs were exported to image software (Adobe Photoshop 3, München, Germany), and two areas were used: one from the wound and another adjacent area. The areas will be compared ( (ΔE) through the Adobe Photoshop red-green chroma scale and the yellow-blue chroma scale according to the following equation: ΔE =[(L.wound- L.adjacent)2 + (a.wound - a.adjacent)2 + (b.wound - b.adjacent)2] 1/ 2 (Knösel et al., 2009).
Epithelialization | 7 days
  It will be analyzed from the percentage of wound epithelialization (% EF) before the surgical procedure and on 7 days thereafter. The wound will be stained with Shirley's solution (Fig. 8) and the epithelial area will be quantified in the Image J. program. Then, with the total area of the wound, the epithelization% will be calculated (Ozcelik et al. 2008).
Tissue thickness | 90 days
  Tissue thickness of palatine masticatory mucosa will be assessed after 90 days of the procedure. For this, an endodontic spacer with a rubber cursor will be put on the donor area for it to reach the palatine bone plate. Then the cursor will be taken to the tissue, not pressuring it. The distance between the spacer tip and the cursor will be measured using a digital paquimeter (Dias et al. 2015).
Postoperative discomfort | 7 days
  Through air spray for 5 s over the operated site, sensitive function will be measured at 7 days after surgical procedure. After air spray application, patients will be required to use a visual analogue scale (VAS) of 100 mm to assess discomfort; scale extremes will be "no pain" to "extreme."
Number of analgesics | 2 weeks
  Patients will be given a postoperative diary in which they will relate the number of analgesics used during 14 days after the procedure. (Tonetti MS et al. 2017).
Tissue edema | 7 days
  Will be evaluated after 7 days of the surgical procedure with the score: 1 = absent; 2 = slight; 3 = moderate; or 4 = severe (Sanz-Molineret, 2013).
Oral Health Impact Profile | 2 weeks
  Will be evaluated from a questionnaire with 14 questions based on 7 domains: functional limitations, physical pain, psychological discomfort, physical disability, psychological deficiency and social deficiency. The patient should respond to the questions within 14 days after the surgical procedure, performing a postoperative diary. For each question an answer must be given, represented in numbers, being: 0- Never; 1- Almost never; 2-Occasionally; 3-Quite frequent; 4-Very common; 5-I do not know (Tonetti MS et al. 2017).

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Principal Investigator — ICT- UNESP
Locations (1):
- Manuela Maria Viana Miguel, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhao M, Penninger J, Isseroff RR. Electrical Activation of Wound-Healing Pathways. Adv Skin Wound Care. 2010 Jan 1;1:567-573. doi: 10.1089/9781934854013.567. PMID 22025904
- [Background] Tomofuji T, Ekuni D, Azuma T, Irie K, Endo Y, Kasuyama K, Nagayama M, Morita M. Effects of electrical stimulation on periodontal tissue remodeling in rats. J Periodontal Res. 2013 Apr;48(2):177-83. doi: 10.1111/j.1600-0765.2012.01518.x. Epub 2012 Aug 14. PMID 22891771